CLINICAL TRIAL: NCT01729923
Title: A Phase II Trial of Maintenance ADAPT Therapy With Capecitabine and Celecoxib in Patients With Metastatic Colorectal Cancer
Brief Title: A Trial of Maintenance ADAPT Therapy With Capecitabine and Celecoxib in Patients With Metastatic Colorectal Cancer
Acronym: ADAPT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stacey Cohen, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7707; NCI-2012-02137 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7707 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Recurrent Colon Carcinoma; Recurrent Rectal Carcinoma; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Celecoxib; Radiotherapy, Intensity-Modulated; Radiotherapy; Radiation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (capecitabine, celecoxib, radiation therapy) (Experimental): Patients proceed to surgery, radiation therapy with ADAPT therapy followed by maintenance ADAPT therapy, or ADAPT therapy. Eligible patients undergo surgical resection at baseline or upon achievement of resectable disease after radiation therapy.
  RADIATION + ADAPT: Patients undergo radiation therapy 5 days per week and receive capecitabine PO BID and celecoxib PO BID 5 days per week during radiation.
  ADAPT: Patients receive capecitabine PO BID on days 1-14 and celecoxib PO BID on days 1-21. Courses repeat every 21 days for up to 3 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Celecoxib; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Radiation: Stereotactic Radiosurgery; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Celecoxib — Given PO
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Radiation: Stereotactic Radiosurgery — Undergo stereotactic radiosurgery
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This phase II trial studies how well capecitabine and celecoxib with or without radiation therapy works in treating patients with colorectal cancer that is newly diagnosed or has been previously treated with fluorouracil, and has spread to other parts of the body (metastatic). Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving capecitabine and celecoxib together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of complete response 2 years following the initiation of first line 5-FU (fluorouracil) based chemotherapy in patients with initially unresected metastatic colorectal cancer who are then treated on the activating cancer stem cells (CSCs) from dormancy and priming them for subsequent targeting (ADAPT) protocol.

SECONDARY OBJECTIVES:

I. To determine overall survival, relapse free survival (if complete response [CR]) based on intent to treat (ITT) analysis.

II. To determine quality of life while on ADAPT therapy.

III. To determine the effects of v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (K-ras) mutation status, resection and radiation on response to ADAPT therapy.

OUTLINE:

Patients proceed to surgery, radiation therapy with ADAPT therapy followed by maintenance ADAPT therapy, or ADAPT therapy. Eligible patients undergo surgical resection at baseline or upon achievement of resectable disease after radiation therapy.

RADIATION + ADAPT: Patients undergo radiation therapy 5 days per week and receive capecitabine orally (PO) twice daily (BID) and celecoxib PO BID 5 days per week during radiation.

ADAPT: Patients receive capecitabine PO BID on days 1-14 and celecoxib PO BID on days 1-21. Courses repeat every 21 days for up to 3 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 2 years, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer
* Evaluable or measurable radiographic evidence of colorectal cancer
* Patients with unresected metastases from colorectal cancer; patients may be either untreated with chemotherapy or currently receiving first-line 5-FU based chemotherapy (folinic acid-fluorouracil-irinotecan hydrochloride [FOLFIRI], capecitabine-irinotecan hydrochloride [CAPIRI], fluorouracil-leucovorin calcium-oxaliplatin [FOLFOX], or capecitabine-oxaliplatin [CAPOX] with or without bevacizumab) within 10 months of beginning ADAPT therapy with at least stable disease radiographically; patients who received prior adjuvant chemotherapy with 5-FU, capecitabine, or FOLFOX are eligible if adjuvant therapy was completed greater than 6 months ago
* History of histological confirmation for recurrent disease, or if recurrent disease is not readily accessible to biopsy, must have two consecutive carcinoembryonic antigen (CEA) or cancer antigen (CA) 19-9 increases, or positron emission tomography (PET) avidity
* Men and women from all ethnic and racial groups
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x the institutional upper-normal limit (IUNL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x IUNL
* Alkaline phosphatase =< 2.5 x IUNL
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,000/uL
* Platelets >= 100,000/uL
* Women of childbearing potential and all men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to beginning ADAPT therapy and for the duration of study participation
* Negative urine pregnancy test for women of childbearing potential
* Must have the ability to understand and the willingness to provide a written informed consent to participate in the study

Exclusion Criteria:

* History of allergies to sulfonamide, aspirin, any nonsteroidal anti-inflammatory drugs (NSAIDS), 5-FU or celecoxib
* Prior 5-FU-based adjuvant chemotherapy less than 6 months prior to beginning ADAPT therapy and any residual neuropathy > grade 2
* Any regular use of cyclooxygenase-2 (COX-2) inhibitors as defined by 2-3 times per week
* Use of aspirin is NOT an exclusion criterion as long as the daily dose does not exceed 325 mg daily; initiation of ADAPT therapy requires patient to discontinue aspirin for 18 months
* Pregnant or lactating women
* History of significant neurologic or psychiatric disorders, including dementia or seizures that would impede consent, treatment, or follow up
* Any serious illness or medical condition that could affect participation on trial
* Any uncontrolled congestive heart failure New York Heart Association class III or IV
* Any uncontrolled hypertension, arrhythmia, or active angina pectoris
* Any history of major myocardial infarction, stroke or transient ischemic attack (TIA); minor acute myocardial infarction (AMI) and patients who have had cardiac bypass free of symptoms for at least 2 years may be eligible at the discretion of the study chair
* Serious uncontrolled active infection
* Patients with creatinine clearance: < 50 mL/min are excluded from this protocol; capecitabine is contraindicated in severe renal impairment (clearance < 40 mL/min)
* Inability to swallow oral medications or any medical conditions that may affect intestinal absorption of the study agent or inability to comply with oral medication
* History of active peptic ulcer disease or major upper gastrointestinal (GI) bleed < 12 months; history of GI bleeding from the colorectal cancer primary is not an exclusion criterion
* Use of warfarin is not allowed; patient is recommended to switch to low molecular weight heparin (LMWH) before participating in this study
* Patients with any history of brain or bone metastasis or who have developed progressive disease on first line 5-FU based therapy
* Current use of systemic steroid medication
* Patients with an obstructive synchronous colorectal tumor requiring up-front surgery or chemoradiation
* Patients with partial or complete bowel obstruction due to abdominal carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09-06 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Cohen, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on March 30, 2013 and terminated on August 12, 2016 due to lack of funding and prior to reaching its enrollment goal. A total 27 participants were accrued.
Groups:
- Treatment (Capecitabine, Celecoxib, Radiation Therapy): Patients proceed to surgery, radiation therapy with ADAPT therapy followed by maintenance ADAPT therapy, or ADAPT therapy. Eligible patients undergo surgical resection at baseline or upon achievement of resectable disease after radiation therapy.
  RADIATION + ADAPT: Patients undergo radiation therapy 5 days per week and receive capecitabine PO BID and celecoxib PO BID 5 days per week during radiation.
  ADAPT: Patients receive capecitabine PO BID on days 1-14 and celecoxib PO BID on days 1-21. Courses repeat every 21 days for up to 3 years in the absence of disease progression or unacceptable toxicity.
  Capecitabine: Given PO
  Celecoxib: Given PO
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
  Radiation Therapy: Undergo radiation therapy
  Stereotactic Radiosurgery: Undergo stereotactic radiosurgery
  Therapeutic Conventional Surgery: Undergo surgical resection
Period: Overall Study
Arm/Group | Treatment (Capecitabine, Celecoxib, Radiation Therapy)
Started | 27
Completed | 0
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Capecitabine, Celecoxib, Radiation Therapy)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 46 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Rate of CR, Assessed According to CEA and CA 19-9 Measurements and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level in response to ADAPT therapy.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Groups:
- Capecitabine and Celecoxib: Patients are treated with oral capecitabine and celecoxib twice daily 7 days per week. Radiation therapy may be used for selected patients. During radiation, treatment with oral capecitabine and celecoxib will be given twice daily 5 days per week. Surgery may also be used for selected patients.
Arm/Group | Capecitabine and Celecoxib
Number analyzed (Participants) | 27
Participants | 1

2. Secondary Outcome: Best Overall Response Rate Among All Patients Who Had RECIST Measurements at Baseline and at Least One Subsequent Occasion
Description: RECIST 1.1 criteria will be used to measure changes in the size of a selected sentinel lesion for each patient. Computed tomographic images will be measured at baseline and at subsequent 9 week intervals. Changes will be measured as percentage of the baseline measure. Results will be reported as the largest negative change. For patients with no negative changes, results will be reported as the smallest positive change.
Time Frame: Serial measures at 9 week intervals up to 5 years
Population: All patients who had RECIST measures at baseline and at least one other time point.
Measure: Mean (Full Range); unit: percentage of baseline lesion size
Arm/Group | Capecitabine and Celecoxib
Number analyzed (Participants) | 19
percentage of baseline lesion size | -17 [-100 to 75.6]

3. Secondary Outcome: Best Overall Response Rate Among All Patients Who Had RECIST Measurements at Baseline and at Least One Subsequent Occasion and Did Not Have Surgery or Radiation Therapy
Description: as for outcome 2
Time Frame: Serial measures at 9 week intervals up to 5 years
Population: Patients who had RECIST measurements at baseline and at least one subsequent occasion and did not have surgery or radiation therapy
Measure: Mean (Full Range); unit: percentage of baseline lesion size
Arm/Group | Capecitabine and Celecoxib
Number analyzed (Participants) | 8
percentage of baseline lesion size | 11 [-31.2 to 75.6]

4. Secondary Outcome: K-ras Mutation Status
Description: The relationship between K-ras mutation, resection, and radiation and response to ADAPT therapy will be evaluated using Chi-squared analysis and Cox regression analysis.
Time Frame: Up to 5 years
Population: K-ras mutation status was not collected.
Arm/Group | Capecitabine and Celecoxib
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method based on the ITT population starting from the time of induction chemotherapy initiation until death or last reported survival.
Time Frame: Until death or last reported survival, up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Capecitabine and Celecoxib
Number analyzed (Participants) | 27
months | 15 [2 to 30]

6. Secondary Outcome: Quality of Life (QOL), Assessed Using the M.D. Anderson Symptom Inventory (MDASI)
Description: Group differences in QOL will be estimated, with repeated measures used to improve precision of estimates.
Time Frame: Up to 5 years
Population: We have been unable to confirmation that the original Principal Investigator secured the appropriate permission to use this instrument. Therefore, we are unable to use the data.
Arm/Group | Capecitabine and Celecoxib
Number analyzed (Participants) | 0

7. Secondary Outcome: Relapse Free Survival in Patients Achieving CR
Description: Relapse-free survival estimated using the Kaplan-Meier method based on the ITT population starting from the time of induction chemotherapy initiation.
Time Frame: Up to 5 years
Population: Measure Description: Inclusive of subject still alive at time of last reporting Time Frame: Until last reported survival Study terminated; data not further analyzed
Measure: Number; unit: months
Arm/Group | Capecitabine and Celecoxib
Number analyzed (Participants) | 1
months | 7

ADVERSE EVENTS:
Time Frame: 3 years
Description: The adverse event recording period will start on the first day of study treatment and end 30 days after last protocol required treatment is administered. Only grade 2 and higher AEs will be recorded with the exception of any AE that requires a dose reduction or treatment interruption.
Arm/Group | Treatment (Capecitabine, Celecoxib, Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 1/27
Other Adverse Events (participants affected / at risk) | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Capecitabine, Celecoxib, Radiation Therapy) (N=27)
Nonoliguric Renal Failure (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Capecitabine, Celecoxib, Radiation Therapy) (N=27)
Diarrhea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 4
Hand/Foot Syndrome (Skin and subcutaneous tissue disorders) | 13
Post-Operative Pain (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 2
Lupus (autoimmune reaction) (Immune system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No